CLINICAL TRIAL: NCT00703326
Title: A Multicenter, Multinational, Randomized, Double-Blind, Phase III Study of IMC-1121B Plus Docetaxel Versus Placebo Plus Docetaxel in Previously Untreated Patients With HER2-Negative, Unresectable, Locally-Recurrent or Metastatic Breast Cancer
Brief Title: Phase III Study of Docetaxel + Ramucirumab or Placebo in Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13892; 2008-001727-65 (EudraCT Number); TRIO-012 (Other: Cancer International Research Group (CIRG)); TRIO-CIRG-012 (Other: Cancer International Research Group (CIRG)); CP12-0606 (Other: ImClone Systems); I4T-IE-JVBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Metastatic breast cancer; HER2 negative breast cancer; locally recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ramucirumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ramucirumab (IMC-1121B) + docetaxel (Experimental)
  Interventions: Biological: ramucirumab (IMC-1121B); Drug: docetaxel
- placebo + docetaxel (Placebo Comparator)
  Interventions: Drug: docetaxel; Other: Placebo

INTERVENTIONS:
Biological: ramucirumab (IMC-1121B) — Ramucirumab (IMC-1121B) is administered at a dose of 10 milligrams per kilogram (mg/kg) as a 1-hour intravenous infusion on Day 1 of each 21-day cycle.
  Other Names: IMC-1121B; LY3009806
  Arms: ramucirumab (IMC-1121B) + docetaxel
Drug: docetaxel — Docetaxel is administered at a dose of 75 milligrams per square meter (mg/m²) as a 1-hour intravenous infusion on Day 1 of each 21-day cycle.
Other: Placebo — Placebo comparator for ramucirumab (IMC-1121B) administered at a dose of 10 mg/kg as a 1-hour intravenous infusion on Day 1 of each 21-day cycle.
  Arms: placebo + docetaxel

SUMMARY:
The objective of this study is to compare the progression-free survival (PFS) of the drug combination ramucirumab plus docetaxel to placebo plus docetaxel in previously untreated participants with human epidermal growth factor receptor 2 (HER2)-negative, unresectable, locally-recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
Female participants at least 18 years of age with histologically or cytologically confirmed, human epidermal growth factor receptor 2 (HER2) negative breast adenocarcinoma that is metastatic or locally-recurrent and inoperable with curative intent will be randomized. Participants may not have received chemotherapy for metastatic or locally-recurrent, inoperable breast cancer.

It is anticipated that 1113 participants will be randomized with 371 participants in the docetaxel plus placebo arm and 742 participants in the docetaxel plus ramucirumab (IMC-1121B) arm. There will be approximately 250 centers in North and South America, Europe, Asia, Middle East, Africa, Australia, and New Zealand.

On Day 1 of each 21-day cycle, participants will receive docetaxel 75 mg/m² as a one-hour I.V. infusion followed by either ramucirumab (IMC-1121B) 10 mg/kg or placebo 10 mg/kg as a one-hour I.V. infusion. Each cycle is repeated every 21 days.

Treatment will continue until there is evidence of progressive disease, unacceptable toxicity, or other withdrawal criteria are met. Participants who discontinue study treatment with either ramucirumab (IMC-1121B) or placebo may continue to receive docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to provide signed informed consent
* Participant is female and ≥ 18 years of age or older if required by local laws or regulations
* Participant has histologically or cytologically confirmed adenocarcinoma of the breast that is now metastatic or locally-recurrent and inoperable with curative intent. Every effort should be made to make paraffin-embedded tissue or slides from the diagnostic biopsy or surgical specimen available for confirmation of diagnosis
* Participant has measurable and/or non-measurable disease
* Participants' primary and/or metastatic tumor is human epidermal growth factor receptor 2 (HER2)-negative by fluorescence in-situ hybridization (FISH) or chromogenic in-situ hybridization (CISH) or 0, 1+ overexpression by immunohistochemistry (IHC)
* Participant has not received prior chemotherapy for metastatic or locally-recurrent and inoperable breast cancer
* Participant completed (neo) adjuvant taxane therapy at least 6 months prior to randomization
* Participant completed (neo) adjuvant biologic therapy at least 6 weeks prior to randomization
* Participant completed all prior radiotherapy with curative intent ≥ 3 weeks prior to randomization
* Participant may have received prior hormonal therapy for breast cancer in the (neo) adjuvant and/or the metastatic setting ≥ 2 weeks prior to randomization
* Participant's left ventricular ejection fraction is within normal institutional ranges
* Participant has resolution to grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3 (NCI-CTCAE v 3.0) of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy with the exception of peripheral neuropathy which must have resolved to grade ≤ 2
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Participant is amenable to compliance with protocol schedules and testing
* Participant has adequate hematological functions [absolute neutrophil count (ANC) ≥ 1500 cells/microliter (mcL), hemoglobin ≥ 9 grams/deciliter (g/dL), and platelets ≥ 100,000 cells/mcL and ≤ 850,000 cells/mcL]
* Participant has adequate hepatic function [bilirubin within normal limits (WNL), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times the upper limit of normal (ULN), or ≤ 5.0 times the ULN if the transaminase elevation is due to liver metastases, and alkaline phosphatase ≤ 5.0 times the ULN]
* Participant has serum creatinine ≤ 1.5 x ULN. If serum creatinine > 1.5 x ULN the calculated creatinine clearance should be > 40 milliliters/minute (mL/min)
* Participant's urinary protein is ≤ 1+ on dipstick or routine urinalysis (UA); if urine protein ≥ 2+, a 24-hour urine collection must demonstrate < 1000 milligrams (mg) of protein in 24 hours to allow participation in the study
* Participant must have adequate coagulation function as defined by international normalized ratio (INR) ≤ 1.5 and a partial thromboplastin time (PTT) ≤ 1.5 X ULN if not receiving anticoagulation therapy. Participants on full-dose anticoagulation must be on a stable dose of oral anticoagulant or low molecular weight heparin and if on warfarin must have a INR between 2 and 3 and have no active bleeding (defined as within 14 days of randomization) or pathological condition that carries a high risk of bleeding (such as, tumor involving major vessels or known varices)
* Women of childbearing potential must implement adequate contraception in the opinion of the investigator
* Participant has not received prior biologic therapy for metastatic or locally recurrent and inoperable breast cancer

Exclusion Criteria:

* Participant has a concurrent active malignancy other than breast adenocarcinoma, adequately treated non melanomatous skin cancer, or other non-invasive carcinoma or in situ neoplasm. A participant with previous history of malignancy is eligible, provided that she has been disease free for > 3 years
* Participant has a known sensitivity to docetaxel or other drugs formulated with polysorbate 80
* Participant has a known sensitivity to agents of similar biologic composition as ramucirumab or other agents that specifically target vascular endothelial growth factor (VEGF)
* Participant has a history of chronic diarrheal disease within 6 months prior to randomization
* Participant has received irradiation to a major bone marrow area as defined as > 25% of bone marrow (such as, pelvic or abdominal radiation) within 30 days prior to randomization
* Participant has participated in clinical trials of experimental agents within 4 weeks prior to randomization
* Participant has a history of uncontrolled hereditary or acquired bleeding or thrombotic disorders
* Participant has active, high risk bleeding (such as, via gastric ulcers or gastric varices) within 14 days prior to randomization
* Participant has an ongoing or active infection requiring parenteral antibiotic, antifungal, or antiviral therapy
* Participant has uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, psychiatric illness/social situations, or any other serious uncontrolled medical disorders in the opinion of the investigator
* Participant has brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease
* Participant has known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness
* Participant has pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
* Participant is pregnant or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1144 (Actual)
Dates: Start 2008-08-06 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (193):
- United States (55):
  - ImClone Investigational Site, Birmingham, Alabama
  - ImClone Investigational Site, Mobile, Alabama
  - ImClone Investigational Site, Chandler, Arizona
  - ImClone Investigational Site, Gilbert, Arizona
  - ImClone Investigational Site, Mesa, Arizona
  - ImClone Investigational Site, Alhambra, California
  - ImClone Investigational Site, Bakersfield, California
  - ImClone Investigational Site, Chula Vista, California
  - ImClone Investigational Site, La Mesa, California
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, Oceanside, California
  - ImClone Investigational Site, Pasadena, California
  - ImClone Investigational Site, San Diego, California
  - ImClone Investigational Site, Santa Barbara, California
  - ImClone Investigational Site, Santa Maria, California
  - ImClone Investigational Site, Santa Monica, California
  - ImClone Investigational Site, Solvang, California
  - ImClone Investigational Site, Valencia, California
  - ImClone Investigational Site, Aurora, Colorado
  - ImClone Investigational Site, Fort Lauderdale, Florida
  - ImClone Investigational Site, Gainesville, Florida
  - ImClone Investigational Site, New Port Richey, Florida
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Macon, Georgia
  - ImClone Investigational Site, Marietta, Georgia
  - ImClone Investigational Site, Alton, Illinois
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Skokie, Illinois
  - ImClone Investigational Site, Elkhart, Indiana
  - ImClone Investigational Site, Mishawaka, Indiana
  - ImClone Investigational Site, South Bend, Indiana
  - ImClone Investigational Site, Westville, Indiana
  - ImClone Investigational Site, Lexington, Kentucky
  - ImClone Investigational Site, Lansing, Michigan
  - ImClone Investigational Site, Saint Joseph, Michigan
  - ImClone Investigational Site, Minneapolis, Minnesota
  - ImClone Investigational Site, Southaven, Mississippi
  - ImClone Investigational Site, St Louis, Missouri
  - ImClone Investigational Site, Grand Island, Nebraska
  - ImClone Investigational Site, Kearney, Nebraska
  - ImClone Investigational Site, Henderson, Nevada
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Charlotte, North Carolina
  - ImClone Investigational Site, Bismarck, North Dakota
  - ImClone Investigational Site, Oklahoma City, Oklahoma
  - ImClone Investigational Site, Portland, Oregon
  - ImClone Investigational Site, West Reading, Pennsylvania
  - ImClone Investigational Site, Bartlett, Tennessee
  - ImClone Investigational Site, Germantown, Tennessee
  - ImClone Investigational Site, Memphis, Tennessee
  - ImClone Investigational Site, Niles, Tennessee
  - ImClone Investigational Site, Oxford, Tennessee
  - ImClone Investigational Site, Lubbock, Texas
  - ImClone Investigational Site, Temple, Texas
  - ImClone Investigational Site, Salt Lake City, Utah
- Australia (19):
  - ImClone Investigational Site, Fitzroy, Victoria
  - ImClone Investigational Site, Frankston, Victoria
  - ImClone Investigational Site, Bankstown
  - ImClone Investigational Site, Bedford Park
  - ImClone Investigational Site, Box Hill
  - ImClone Investigational Site, Darlinghurst
  - ImClone Investigational Site, East Bentleigh
  - ImClone Investigational Site, East Melbourne
  - ImClone Investigational Site, Herston
  - ImClone Investigational Site, Hobart
  - ImClone Investigational Site, Milton
  - ImClone Investigational Site, Nambour
  - ImClone Investigational Site, New Lambton Heights
  - ImClone Investigational Site, Perth
  - ImClone Investigational Site, Ringwood East
  - ImClone Investigational Site, Subiaco
  - ImClone Investigational Site, Sydney
  - ImClone Investigational Site, Tweed Heads
  - ImClone Investigational Site, Wendouree
- Belgium (8):
  - ImClone Investigational Site, Brasschaat
  - ImClone Investigational Site, Charleroi
  - ImClone Investigational Site, Edegem
  - ImClone Investigational Site, Ghent
  - ImClone Investigational Site, Kortrijk
  - ImClone Investigational Site, Liège
  - ImClone Investigational Site, Namur
  - ImClone Investigational Site, Yvoir
- Brazil (5):
  - ImClone Investigational Site, Ijuí
  - ImClone Investigational Site, Porto Alegre
  - ImClone Investigational Site, Rio de Janeiro
  - ImClone Investigational Site, Santo André
  - ImClone Investigational Site, São Paulo
- Canada (7):
  - ImClone Investigational Site, Calgary, Alberta
  - ImClone Investigational Site, Edmonton, Alberta
  - ImClone Investigational Site, Vancouver, British Columbia
  - ImClone Investigational Site, Toronto, Ontario
  - ImClone Investigational Site, Weston, Ontario
  - ImClone Investigational Site, Greenfield Park, Quebec
  - ImClone Investigational Site, Québec
- ImClone Investigational Site, Osijek, Croatia
- Czechia (6):
  - ImClone Investigational Site, Prague, Motol
  - ImClone Investigational Site, Brno
  - ImClone Investigational Site, Kutná Hora
  - ImClone Investigational Site, Pardubice
  - ImClone Investigational Site, Prague
  - ImClone Investigational Site, Videnska
- Egypt (2):
  - ImClone Investigational Site, Alexandria
  - ImClone Investigational Site, Cairo
- Germany (10):
  - ImClone Investigational Site, Chemnitz
  - ImClone Investigational Site, Hamburg
  - ImClone Investigational Site, Kiel
  - ImClone Investigational Site, Lübeck
  - ImClone Investigational Site, Munich
  - ImClone Investigational Site, München
  - ImClone Investigational Site, Oldenburg
  - ImClone Investigational Site, Saarbrücken
  - ImClone Investigational Site, Trier
  - ImClone Investigational Site, Tübingen
- Ireland (4):
  - ImClone Investigational Site, Cork
  - ImClone Investigational Site, Dublin
  - ImClone Investigational Site, Erlangen
  - ImClone Investigational Site, Limerick
- Israel (5):
  - ImClone Investigational Site, Beersheva
  - ImClone Investigational Site, Jerusalem
  - ImClone Investigational Site, Petah Tikva
  - ImClone Investigational Site, Rehovot
  - ImClone Investigational Site, Tel Aviv
- Lebanon (5):
  - ImClone Investigational Site, Beirut
  - ImClone Investigational Site, Bsalîm
  - ImClone Investigational Site, Metn
  - ImClone Investigational Site, Sidon
  - ImClone Investigational Site, Zghartā
- New Zealand (2):
  - ImClone Investigational Site, Auckland
  - ImClone Investigational Site, Palmerston North
- Peru (2):
  - ImClone Investigational Site, Arequipa
  - ImClone Investigational Site, Lima
- Poland (2):
  - ImClone Investigational Site, Bytom
  - ImClone Investigational Site, Olsztyn
- Russia (16):
  - ImClone Investigational Site, Engel's
  - ImClone Investigational Site, Kazan'
  - ImClone Investigational Site, Kursk
  - ImClone Investigational Site, Leningrad Region
  - ImClone Investigational Site, Lipetsk
  - ImClone Investigational Site, Magnitogorsk
  - ImClone Investigational Site, Moscow
  - ImClone Investigational Site, Novosibirsk
  - ImClone Investigational Site, Omsk
  - ImClone Investigational Site, Orenburg
  - ImClone Investigational Site, Perm
  - ImClone Investigational Site, Saint Petersburg
  - ImClone Investigational Site, Samara
  - ImClone Investigational Site, Saratov
  - ImClone Investigational Site, Tambov
  - ImClone Investigational Site, Ufa
- Serbia (3):
  - ImClone Investigational Site, Kamenitz
  - ImClone Investigational Site, Kragujevac
  - ImClone Investigational Site, Niš
- Slovakia (3):
  - ImClone Investigational Site, Bratislava
  - ImClone Investigational Site, Trnava
  - ImClone Investigational Site, Žilina
- South Africa (8):
  - ImClone Investigational Site, Parktown, Johannesburg
  - ImClone Investigational Site, Bloemfontein
  - ImClone Investigational Site, Durban
  - ImClone Investigational Site, eManzimtoti
  - ImClone Investigational Site, Lynnwood
  - ImClone Investigational Site, Port Elizabeth
  - ImClone Investigational Site, Pretoria
  - ImClone Investigational Site, Sandton
- South Korea (2):
  - ImClone Investigational Site, Incheon
  - ImClone Investigational Site, Seoul
- Spain (19):
  - ImClone Investigational Site, A Coruña
  - ImClone Investigational Site, Alicante
  - ImClone Investigational Site, Badalona
  - ImClone Investigational Site, Barbastro
  - ImClone Investigational Site, Barcelona
  - ImClone Investigational Site, Donostia / San Sebastian
  - ImClone Investigational Site, Girona
  - ImClone Investigational Site, Jaén
  - ImClone Investigational Site, La Laguna - Tenerife
  - ImClone Investigational Site, Lleida
  - ImClone Investigational Site, Madrid
  - ImClone Investigational Site, Málaga
  - ImClone Investigational Site, Palma de Mallorca
  - ImClone Investigational Site, Salamanca
  - ImClone Investigational Site, Santander
  - ImClone Investigational Site, Seville
  - ImClone Investigational Site, Toledo
  - ImClone Investigational Site, Valencia
  - ImClone Investigational Site, Zaragoza
- Taiwan (3):
  - ImClone Investigational Site, Changhua
  - ImClone Investigational Site, Taipei
  - ImClone Investigational Site, Taoyuan
- United Kingdom (6):
  - ImClone Investigational Site, Bournemouth
  - ImClone Investigational Site, Edinburgh
  - ImClone Investigational Site, Huddersfield
  - ImClone Investigational Site, Hull
  - ImClone Investigational Site, Manchester
  - ImClone Investigational Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and european union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org

REFERENCES:
- [Derived] Arnold D, Fuchs CS, Tabernero J, Ohtsu A, Zhu AX, Garon EB, Mackey JR, Paz-Ares L, Baron AD, Okusaka T, Yoshino T, Yoon HH, Das M, Ferry D, Zhang Y, Lin Y, Binder P, Sashegyi A, Chau I. Meta-analysis of individual patient safety data from six randomized, placebo-controlled trials with the antiangiogenic VEGFR2-binding monoclonal antibody ramucirumab. Ann Oncol. 2017 Dec 1;28(12):2932-2942. doi: 10.1093/annonc/mdx514. PMID 28950290
- [Derived] Spera G, Fresco R, Fung H, Dyck JRB, Pituskin E, Paterson I, Mackey JR. Beta blockers and improved progression-free survival in patients with advanced HER2 negative breast cancer: a retrospective analysis of the ROSE/TRIO-012 study. Ann Oncol. 2017 Aug 1;28(8):1836-1841. doi: 10.1093/annonc/mdx264. PMID 28520849
- [Derived] Mackey JR, Ramos-Vazquez M, Lipatov O, McCarthy N, Krasnozhon D, Semiglazov V, Manikhas A, Gelmon KA, Konecny GE, Webster M, Hegg R, Verma S, Gorbunova V, Abi Gerges D, Thireau F, Fung H, Simms L, Buyse M, Ibrahim A, Martin M. Primary results of ROSE/TRIO-12, a randomized placebo-controlled phase III trial evaluating the addition of ramucirumab to first-line docetaxel chemotherapy in metastatic breast cancer. J Clin Oncol. 2015 Jan 10;33(2):141-8. doi: 10.1200/JCO.2014.57.1513. Epub 2014 Sep 2. PMID 25185099

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were alive and completed the follow-up period or who died were considered to have completed the study.
Groups:
- Ramucirumab (IMC-1121B) + Docetaxel: Ramucirumab (IMC-1121B) is administered at a dose of 10 milligrams per kilogram (mg/kg) as a 1-hour intravenous infusion on Day 1 of each 21-day cycle.
  Docetaxel is administered at a dose of 75 milligrams per square meter (mg/m²) as a 1-hour intravenous infusion on Day 1 of each 21-day cycle.
- Placebo + Docetaxel: Placebo comparator for ramucirumab (IMC-1121B) administered at a dose of 10 mg/kg as a 1-hour intravenous infusion on Day 1 of each 21-day cycle.
  Docetaxel is administered at a dose of 75 milligrams per square meter (mg/m²) as a 1-hour intravenous infusion on Day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel
Started | 759 | 385
Received at Least 1 Dose of Study Drug | 752 | 382
Completed | 657 | 347
Not Completed | 102 | 38
Not completed — Lost to Follow-up | 47 | 18
Not completed — Withdrawal by Subject | 54 | 20
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel | Total
Number analyzed (Participants) | 759 | 385 | 1144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 629 | 325 | 954
  >=65 years | 130 | 60 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.5) | 54.2 (10.0) | 54.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 759 | 385 | 1144
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69 | 42 | 111
  Not Hispanic or Latino | 690 | 343 | 1033
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 31 | 20 | 51
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 27 | 14 | 41
  White | 676 | 341 | 1017
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 9 | 31
Region of Enrollment [Count of Participants; unit: Participants]
  Serbia | 0 | 2 | 2
  United States | 58 | 21 | 79
  Taiwan | 4 | 2 | 6
  Slovakia | 2 | 2 | 4
  Spain | 118 | 64 | 182
  Lebanon | 24 | 14 | 38
  Ireland | 8 | 2 | 10
  Russia | 210 | 99 | 309
  Israel | 16 | 7 | 23
  United Kingdom | 21 | 10 | 31
  Egypt | 9 | 3 | 12
  Czechia | 4 | 3 | 7
  Canada | 83 | 46 | 129
  Poland | 12 | 5 | 17
  Belgium | 48 | 20 | 68
  Brazil | 30 | 20 | 50
  Peru | 12 | 4 | 16
  Australia | 28 | 21 | 49
  South Africa | 41 | 22 | 63
  Germany | 12 | 5 | 17
  New Zealand | 5 | 6 | 11
  South Korea | 14 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as time from randomization until the first evidence of progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.0) or death from any cause; by Investigator assessment. Progressive disease (PD) was defined as at least a 20% increase in sum of longest diameter of target lesions taking as reference the smallest sum longest diameter since baseline, progression in non-target lesions or the appearance of 1 or more new lesion(s). Participants who neither progressed nor died were censored the day of their last radiographic tumor assessment if available or date of randomization if no post initiation radiographic assessment was available. If death or PD occurred after ≥2 missing radiographic visits, censoring occurred at date of the last radiographic visit prior to the missed visits. The symptomatic/clinical disease progression (deterioration) without documented radiologic progression did not constitute progression.
Time Frame: Randomization to disease progression or death or until data cutoff of 31 Mar 2013 (up to 56 months)
Population: Intent-to-Treat (ITT) Population: All randomized participants. Censored participants: ramucirumab + docetaxel=231, placebo + docetaxel=94.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 759 | 385
months | 9.5 [8.3 to 9.8] | 8.2 [7.1 to 8.5]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1121B) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.077, Stratified Log Rank (SLR); SLR used Interactive Web Response System (IWRS) factors: prior taxane therapy, visceral metastasis, hormone receptor status and geographical regions; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.75 to 1.01] — HR with 95% confidence interval (CI) was estimated using a stratified Cox proportional hazards regression model using the IWRS stratification factors

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from randomization to death from any cause. Participants who were alive at data cut-off for the OS analysis or lost to follow-up were censored on the last date the participant was known to be alive.
Time Frame: Randomization to death or until data cutoff of 29-May-2015 (up to 82 months)
Population: Intent-to-Treat (ITT) Population: All randomized participants. Censored participants: ramucirumab + docetaxel=267, placebo + docetaxel=121.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 759 | 385
months | 30.3 [27.5 to 33.5] | 28.7 [25.6 to 32.3]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1121B) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.487, Stratified Log Rank (SLR) — The gate-keeping strategy used to control overall type 1 error 0.05 (2-sided) or 0.025 (1-sided) to analyze progression-free survival (PFS) and OS. At final PFS analysis only if primary PFS test was significant would analysis of OS be inferential; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.81 to 1.10] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from the date of randomization to the first documented date of disease progression using Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria; by Investigator assessment. Progressive disease (PD) was defined as at least a 20% increase in sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD since baseline, progression in non-target lesions or the appearance of 1 or more new lesion(s). Participants who did not progress were censored at the last radiographic tumor assessment. If no post-baseline assessment was available censoring occurred at the date of randomization. If PD occurred after 2 or more missing radiographic visits, censoring occurred at the date of the last radiographic visit prior to the missed visits. The symptomatic/clinical disease progression (deterioration) without documented radiologic progression did not constitute progression.
Time Frame: Randomization to disease progression or until data cutoff of 31-Mar-2013 (up to 56 months)
Population: Intent-to-Treat (ITT) Population: All randomized participants. Censored participants: ramucirumab + docetaxel=263, placebo + docetaxel=104.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 759 | 385
months | 9.7 [8.5 to 10.3] | 8.2 [7.1 to 9.0]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1121B) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.033, Stratified Log Rank (SLR); [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.73 to 0.99] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate)
Description: Objective response rate (ORR) was defined as the percentage of randomized participants achieving a best confirmed overall response of CR or PR using Response Evaluation Criteria in Solid Tumors (RECIST v1.0), based on the achievement of both measurement and confirmation criteria; by Investigator assessment. CR was defined as the disappearance of all target and non-target lesions. PR was defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions, taking as reference the baseline sum LD and no progression in non-target lesions.
Time Frame: Randomization to disease progression or until data cutoff of 31-Mar-2013 (up to 56 months)
Population: Intent-to-Treat (ITT) Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 759 | 385
percentage of participants | 44.7 [41.1 to 48.3] | 37.9 [33.1 to 43.0]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1121B) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.027, Stratified Cochran-Mantel-Haenszel(SCMH); SCMH used Interactive Web Response System (IWRS) factors: prior taxane therapy, visceral metastasis, hormone receptor status and geographical regions; Odds Ratio (OR) = 1.33, 95% CI 2-sided [1.03 to 1.71] — Stratified odds ratio was calculated considering the IWRS stratification factors

5. Secondary Outcome: Duration of Response
Description: Duration of complete response (CR) or partial response (PR) measured from time criteria were first met for CR or PR until first date of progressive disease (PD) or death from any cause defined using Response Evaluation Criteria in Solid Tumor (RECIST 1.0); by Investigator assessment. CR defined as disappearance of all target and non-target lesions. PR defined as ≥30% decrease in sum of longest diameter (LD) of target lesions and no progression in non-target lesions. PD defined as ≥20% increase in LD sum of target lesions taking as reference the smallest sum LD since baseline, progression in non-target lesions or the appearance of ≥1 new lesion(s). Participants who did not relapse or die censored at day of last radiographic tumor assessment. If death or PD was after ≥2 missing radiographic visits, censoring was at date of last radiographic visit prior to missed visits. Symptomatic/clinical disease progression without documented radiologic progression did not constitute progression.
Time Frame: Date of first CR or PR to PD or death or until data cutoff date of 31-Mar-2013 (up to 56 months)
Population: A subset of the Intent-to-Treat (ITT) Population: all randomized participants with CR or PR. Censored participants: ramucirumab + docetaxel=80, placebo + docetaxel=28.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 339 | 146
months | 8.4 [8.0 to 9.7] | 8.1 [6.8 to 8.9]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1121B) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.150, Stratified Log Rank (SLR); [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.67 to 1.06] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Total Functional Assessment of Cancer Therapy-Breast (FACT-B): Change From Baseline to End of Therapy
Description: FACT-B measures the following domains of health-related quality of life (HR-QoL): physical well-being (PWB), social/family well-being (SFWB), emotional well-being (EWB), functional well-being (FWB), and additional concerns of breast cancer subscale (BCS) each with 6 or more items developed to measure problems specific to breast cancer symptoms plus additional items related to global QoL. Participants respond to each of the 36 questions on a 5-point scale from 0 (not at all) to 4 (very much) with a total scores range of 0-144. Higher scores indicate fewer symptoms and better HR-QoL.
Time Frame: Baseline, End of Therapy or until data cutoff of 31-Mar-2013 (up to 56 months)
Population: A subset of Intent-to-Treat (ITT) Population: all randomized participants with a valid baseline and end of therapy assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 494 | 251
units on a scale | -6.8 (17.3) | -7.0 (16.8)
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1121B) + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.539, ANCOVA — P-value is for end of therapy. Analysis of covariance (ANCOVA) adjusted for baseline score was used to compare the 2 treatment arms

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Clinically significant events were defined as serious adverse events (SAE) and other treatment-emergent non-serious adverse events (NSAE). A summary of SAEs and other NSAEs is located in the Reported Adverse Event module.
Time Frame: First dose to study completion (up to 12.3 years)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 752 | 382
participants
  Participants with SAEs | 285 | 117
  Participants with NSAEs | 737 | 373

8. Secondary Outcome: Immunogenicity: Percentage of Participants With Treatment Emergent Anti-Ramucirumab Antibodies Until Primary Data Cutoff of 31-Mar-2013
Description: Percentage of participants with treatment-emergent positive for anti-ramucirumab (IMC-1121B) antibodies during the study. Participants were considered positive for anti-ramucirumab (IMC-1121B) antibodies if they exhibited a post-treatment antibody level that exceeded the positive upper cut point determined from the anti-ramucirumab (IMC-1121B) level seen in healthy untreated individuals.
Time Frame: Baseline, prior to cycle 3 infusion, prior to cycle 5 infusion, onset of infusion reaction, resolution of reaction and 30 days following the event up to 56 months
Population: All randomized participants who received at least 1 dose of study drug with anti-IMC-1121B antibodies samples collected during the study.
Measure: Number; unit: percentage of participants
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 715 | 360
percentage of participants | 0.8 | 0.8

9. Secondary Outcome: Immunogenicity: Percentage of Participants Available After 31-Mar-2013 With Treatment Emergent Anti-Ramucirumab Antibodies Until Data Cutoff From 01-Apr-2013 to 08-Sep-2016
Description: as for outcome 8
Time Frame: Follow-up from 01-Apr-2013 to 08-Sep-2016 (Up to 56 -97 months)
Population: All follow-up participants (additional participants who were available after primary data cut off 31-Mar-13) who received at least 1 dose of study drug with anti-IMC-1121B antibodies samples collected during the study.
Measure: Number; unit: percentage of participants
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 35 | 22
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose to study completion (up to 12.3 years)
Description: All randomized participants who received at least 1 dose of study drug. Disease progression without clinical manifestation or death related to progressive disease (PD) was not to be reported as an adverse event (AE). However, all deaths within 30 days of last dose were reported as a serious AE (SAE), regardless of causality. PD itself was reported as an SAE, if any of the SAE criteria were met.
Arm/Group | Ramucirumab (IMC-1121B) + Docetaxel | Placebo + Docetaxel
Serious Adverse Events (participants affected / at risk) | 285/752 | 117/382
Other Adverse Events (participants affected / at risk) | 737/752 | 373/382
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (IMC-1121B) + Docetaxel (N=752) | Placebo + Docetaxel (N=382)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 51 (57) | 11 (12)
Neutropenia (Blood and lymphatic system disorders) | 47 (52) | 20 (23)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (3) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Panophthalmitis (Eye disorders) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 2 (2)
Diverticular perforation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 9 (11) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (7) | 2 (2)
Asthenia (General disorders) | 5 (5) | 1 (1)
Chills (General disorders) | 3 (3) | 0 (0)
Complication associated with device (General disorders) | 2 (2) | 2 (2)
Death (General disorders) | 2 (2) | 0 (0)
Disease progression (General disorders) | 8 (8) | 4 (4)
Extravasation (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 10 (10) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 1 (1)
Generalised oedema (General disorders) | 2 (2) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0)
Infusion site thrombosis (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 8 (9) | 2 (2)
Sudden death (General disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 4 (5) | 3 (3)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Abscess soft tissue (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Anal infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 8 (8) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 4 (4) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic infection (Infections and infestations) | 19 (19) | 9 (10)
Neutropenic sepsis (Infections and infestations) | 7 (7) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 15 (16) | 5 (5)
Pneumonia chlamydial (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (7) | 3 (3)
Vascular device infection (Infections and infestations) | 4 (6) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical burn of skin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Expired product administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 9 (9) | 2 (2)
Overdose (Injury, poisoning and procedural complications) | 7 (13) | 5 (11)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Product administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Product dispensing error (Injury, poisoning and procedural complications) | 3 (3) | 1 (2)
Product preparation issue (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Underdose (Injury, poisoning and procedural complications) | 11 (34) | 12 (24)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrong product administered (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (8) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (2) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 4 (4) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Disability (Social circumstances) | 0 (0) | 1 (1)
Therapy change (Surgical and medical procedures) | 0 (0) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 3 (3)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 2 (2)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (IMC-1121B) + Docetaxel (N=752) | Placebo + Docetaxel (N=382)
Anaemia (Blood and lymphatic system disorders) | 77 (108) | 28 (39)
Neutropenia (Blood and lymphatic system disorders) | 96 (175) | 41 (56)
Tachycardia (Cardiac disorders) | 50 (70) | 23 (36)
Lacrimation increased (Eye disorders) | 233 (337) | 65 (90)
Abdominal pain (Gastrointestinal disorders) | 95 (141) | 42 (59)
Abdominal pain upper (Gastrointestinal disorders) | 51 (71) | 24 (33)
Constipation (Gastrointestinal disorders) | 157 (293) | 74 (116)
Diarrhoea (Gastrointestinal disorders) | 326 (751) | 152 (338)
Dry mouth (Gastrointestinal disorders) | 29 (54) | 20 (33)
Dyspepsia (Gastrointestinal disorders) | 75 (110) | 40 (57)
Gingival bleeding (Gastrointestinal disorders) | 73 (144) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 39 (50) | 8 (8)
Nausea (Gastrointestinal disorders) | 278 (766) | 156 (343)
Stomatitis (Gastrointestinal disorders) | 380 (833) | 118 (215)
Vomiting (Gastrointestinal disorders) | 155 (288) | 80 (127)
Asthenia (General disorders) | 270 (549) | 127 (363)
Face oedema (General disorders) | 73 (100) | 27 (30)
Fatigue (General disorders) | 271 (481) | 135 (240)
Influenza like illness (General disorders) | 39 (48) | 29 (40)
Non-cardiac chest pain (General disorders) | 39 (43) | 19 (21)
Oedema (General disorders) | 43 (48) | 18 (26)
Oedema peripheral (General disorders) | 181 (274) | 101 (140)
Pyrexia (General disorders) | 110 (168) | 44 (65)
Conjunctivitis (Infections and infestations) | 38 (42) | 17 (25)
Nasopharyngitis (Infections and infestations) | 63 (79) | 20 (30)
Upper respiratory tract infection (Infections and infestations) | 39 (48) | 21 (29)
Urinary tract infection (Infections and infestations) | 71 (91) | 28 (32)
Infusion related reaction (Injury, poisoning and procedural complications) | 41 (56) | 24 (43)
Weight decreased (Investigations) | 173 (209) | 41 (50)
Weight increased (Investigations) | 123 (152) | 92 (105)
Decreased appetite (Metabolism and nutrition disorders) | 165 (293) | 62 (101)
Arthralgia (Musculoskeletal and connective tissue disorders) | 173 (359) | 82 (167)
Back pain (Musculoskeletal and connective tissue disorders) | 114 (143) | 54 (74)
Bone pain (Musculoskeletal and connective tissue disorders) | 92 (192) | 41 (82)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 51 (105) | 18 (32)
Myalgia (Musculoskeletal and connective tissue disorders) | 153 (292) | 89 (209)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 107 (195) | 47 (66)
Dizziness (Nervous system disorders) | 64 (88) | 36 (45)
Dysgeusia (Nervous system disorders) | 68 (120) | 32 (66)
Headache (Nervous system disorders) | 171 (306) | 70 (98)
Neuropathy peripheral (Nervous system disorders) | 101 (124) | 64 (78)
Paraesthesia (Nervous system disorders) | 47 (59) | 31 (40)
Peripheral sensory neuropathy (Nervous system disorders) | 136 (193) | 73 (90)
Taste disorder (Nervous system disorders) | 105 (156) | 58 (89)
Anxiety (Psychiatric disorders) | 49 (65) | 27 (27)
Insomnia (Psychiatric disorders) | 99 (127) | 33 (39)
Proteinuria (Renal and urinary disorders) | 44 (75) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 127 (179) | 69 (89)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 163 (225) | 75 (90)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 300 (817) | 64 (149)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 65 (96) | 27 (36)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 69 (74) | 28 (29)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 56 (82) | 19 (23)
Alopecia (Skin and subcutaneous tissue disorders) | 535 (550) | 279 (287)
Dry skin (Skin and subcutaneous tissue disorders) | 55 (60) | 21 (21)
Nail disorder (Skin and subcutaneous tissue disorders) | 231 (250) | 105 (114)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 106 (157) | 33 (36)
Pruritus (Skin and subcutaneous tissue disorders) | 41 (44) | 21 (23)
Rash (Skin and subcutaneous tissue disorders) | 109 (143) | 47 (63)
Hot flush (Vascular disorders) | 34 (44) | 21 (22)
Hypertension (Vascular disorders) | 204 (405) | 44 (96)

LIMITATIONS AND CAVEATS:
One participant assigned to placebo + docetaxel (doc) treatment and was given ramucirumab (ram) in Cycle 1. Considered ram + doc treatment arm for safety population, for ITT population the participant was analyzed according to assigned treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.